CLINICAL TRIAL: NCT01264211
Title: A 6-month Pilot Randomised Double-blind Placebo-controlled Multicentre, Phase 2 Study
Brief Title: Safety and Efficacy of the Combination of Diacerein 100 mg Daily and MTX Versus MTX Alone in the Treatment of Early Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TRB Chemedica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAR-THA-05-01
Record Dates: First submitted 2010-06-28; First posted 2010-12-21 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Efficacy of Diacerein; Safety of Diacerein; Carry-over effect of Diacerein
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — diacerein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diacerein (Experimental)
  Interventions: Drug: Diacerein
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diacerein — Week 0 to Week 4: Diacerein 50 mg daily for 4 weeks Week 4 to Week 24: Diacerein 100 mg daily for 20 weeks
  Arms: Diacerein
Drug: Placebo — Week 0 to Week 4: Diacerein 50 mg daily for 4 weeks Week 4 to Week 24: Diacerein 100 mg daily for 20 weeks
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of Diacerein 100 mg daily versus placebo in reducing rheumatoid arthritis symptoms, when added to stable oral MTX therapy in patients with active early RA.

To evaluate the safety of Diacerein 100 mg daily when administrated in combination with oral MTX therapy in those patients for up to 24 weeks

To investigate a potential persistent effect, 4 weeks after Diacerein treatment is stopped (carry-over effect)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18 and 65 years;
2. Active RA of ≥ 3 months duration but < 2 years, diagnosed according to the American College of Rheumatology (ACR) 1987 revised criteria for RA;
3. RA global functional status class I-III;
4. Treatment on an outpatient basis;
5. Treatment with MTX for a minimum of 12 weeks, with stable weekly dose (10-20 mg) for at least 4 weeks before randomisation;
6. Insufficient response to treatment with MTX, with disease activity score DAS28 > 4.0 at the time of screening and randomisation; the DAS28 must not change significantly from screening to baseline visit (change < 0.6);
7. Tender joint count (TJC) ≥ 6 (68 joint count) and swollen joint count (SJC) ≥ 6 (66 joint count) at screening and randomisation;
8. Screening ESR ≥ 28 mm/h;
9. Evidence of adequate contraceptive methods in women of childbearing potential. Female patients of childbearing potential are those who are not surgically sterile or post-menopausal. Adequate contraceptive methods are hormonal contraceptive, intra-uterine device, diaphragm with spermicide or condom with spermicide for the entire duration of the study;
10. Agreement not to drink alcohol for the duration of the study;
11. Ability and agreement to comply with the requirements of the study protocol;
12. Having given written informed consent to participate in the study.

Exclusion Criteria:

1. History of active inflammatory arthritis other than RA;
2. Any uncontrolled medical condition such as diabetes mellitus, asthma, cardiopulmonary disease, congestive heart failure, neurological disease, etc.;
3. Alcohol abuse, defined as the consumption of more than one glass of beer or wine in a day;
4. Moderate or severe liver disease (cirrhosis, hepatitis, liver insufficiency);
5. Blood anomalies (significant cytopenia);
6. History of, or currently active primary or secondary immunodeficiency;
7. Chronic hepatitis B (HBsAg positive or HBcAb positive with HBV DNA load ≥ 400 copies/ml) or hepatitis C (anti-HCV positive);
8. Current known active, or history of, recurrent bacterial, viral, fungal, mycobacterial or other infections, or any infection requiring hospitalisation or treatment with i.v. antibiotics within 4 weeks prior to randomisation or oral antibiotics within 2 weeks prior to randomisation;
9. Treatment with biologic DMARDs such as TNF antagonists, IL 1 receptor antagonists, IL 6 receptor antagonists, CTLA4Ig within 12 weeks prior to randomisation, and rituximab within 24 weeks prior to randomisation;
10. Treatment with non-biologic DMARDs such as chloroquine, hydroxychloroquine, penicillamine, sulfasalazine within 4 weeks prior to randomisation, leflunomide, parenteral gold, oral gold within 8 weeks prior to randomisation, azathioprine and ciclosporin within 12 weeks prior to randomisation;
11. Treatment with intra-articular injection of a depocorticosteroid within 8 weeks prior to randomisation;
12. Treatment with NSAID or oral corticosteroids, unless the patient has been on a stable dose for at least 4 weeks before randomisation (maximal allowed daily dose of oral corticosteroid equivalent to prednisone 10 mg);
13. Physical therapy and alternative therapies, unless the patient has received them regularly for at least 4 weeks before randomisation;
14. Initiation of chronic treatment with antihistaminics, antidepressants or tranquilisers, within less than 12 weeks before randomisation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with ACR20 response criteria | 24 weeks

SECONDARY OUTCOMES:
Percentage of patients achieving a moderate response according to EULAR response criteria (changes in DAS28 score) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Juree Rawdmanee, Sukhumvit, Bangkok
  - Faculty of medicine, Chiangmai University, Chiang Mai, Chiangmai

REFERENCES:
- [Derived] Louthrenoo W, Nilganuwong S, Nanagara R, Siripaitoon B, Collaud Basset S. Diacerein for the treatment of rheumatoid arthritis in patients with inadequate response to methotrexate: a pilot randomized, double-blind, placebo-controlled add-on trial. Clin Rheumatol. 2019 Sep;38(9):2461-2471. doi: 10.1007/s10067-019-04587-1. Epub 2019 May 19. PMID 31104217